CLINICAL TRIAL: NCT00628901
Title: A Prospective, Randomized, Single-Center Study Comparing Contour SE™ Microspheres to Embosphere® Microspheres for Treating Symptomatic Uterine Fibroids With Uterine Fibroid Embolization (UFE)
Brief Title: A Prospective Study Comparing Contour SE™ Microspheres to Embosphere® Microspheres for Treating Symptomatic Uterine Fibroids With Uterine Fibroid Embolization (UFE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M9011; ONC-PM-022005
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2011-08-22 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Leiomyoma; Uterine Fibroids; Uterine Neoplasms; Menorrhagia; Leiomyomatosis
Keywords: Leiomyoma; Uterine Fibroids; Uterine Fibroid Embolization (UFE); Uterine Artery Embolization (UAE); Uterine Neoplasms; Menorrhagia
MeSH Terms: conditions — Leiomyoma; Uterine Neoplasms; Menorrhagia; Leiomyomatosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Procedure: Uterine Fibroid Embolization (UFE); Device: Contour SE™ Microspheres
- Arm 2 (Active Comparator)
  Interventions: Procedure: Uterine Fibroid Embolization (UFE); Device: Embosphere® Microspheres

INTERVENTIONS:
Procedure: Uterine Fibroid Embolization (UFE) — Uterine Fibroid Embolization is used in treating Uterine Fibroids. The procedure involves injecting embolization particles into the fibroid via the uterine artery which causes the fibroid to shrink or subside. Patients are usually released from the hospital the day after the procedure.
Device: Contour SE™ Microspheres — Polyvinyl alcohol Microsphere embolization devices intended to provide targeted vascular occlusion or reduction of blood flow upon selective placement and are currently marketed for use in hypervascular tumors, including leiomyoma uteri and arteriovenous malformations
  Arms: Arm 1
Device: Embosphere® Microspheres — Biocompatible, hydrophilic, nonresorbable, microspheres used in the embolization of arteriovenous malformations, hypervascular tumors, and symptomatic uterine fibroids.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to demonstrate comparability between Contour SE™ Microspheres and Embosphere® Microspheres for achieving post UFE fibroid devascularization in women with symptomatic uterine fibroids.

DETAILED DESCRIPTION:
The purpose of this prospective randomized single-center study is to demonstrate comparability using Contour SE™ Microspheres (700-900µ and 900-1200µ) using a near stasis endpoint and Embosphere® Microspheres (500-700µ) using a "prune tree" endpoint for achieving post UFE fibroid devascularization in women with symptomatic uterine fibroids. The study will demonstrate (with the use of contrast enhanced Magnetic Resonance Imaging (MRI) at baseline and 24-hours post embolization) that uterine fibroids can successfully be devascularized using the embolization protocols. Contrast enhanced MRI will be performed at baseline, 24-hours, and 3-months post UFE. The subjects will be followed through 12-months post UFE and change from baseline in symptom severity (Quality of Life (QoL) Questionnaire) will be assessed at 3 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the following symptoms: abnormal menstrual bleeding, infertility related to fibroids, pelvic pain, and/or bulk/pressure related symptoms attributed to fibroids: i.e., pelvic pressure, abdominal enlargement, abdominal bloating, gastrointestinal pressure symptoms (backache, constipation), dysfunction of the urinary bladder (urinary frequency, urinary retention), vaginal pressure, and rectal pressure.
* Severity of the symptom(s) warrants invasive treatment
* Willing and able to complete the follow-up requirements outlined in the study design section of the protocol
* Willing to sign a consent form

Exclusion Criteria:

* Active pelvic inflammatory disease or infection
* Any malignancy of the pelvic region
* Endometrial neoplasia or hyperplasia
* Presence of one or more submucosal fibroid(s) with more than 50% growth into the uterine cavity
* Presence of pedunculated serosal fibroid as the dominant fibroid(s)
* Fibroids with significant collateral feeding by vessels other than the uterine arteries
* Presence of arteries supplying the fibroid are not large enough to accept 700-900 micron or 900-1200 micron microspheres
* Coagulopathy
* Atypical anatomy that will not allow for bilateral UFE
* Subject with known severe contrast allergy
* Subjects with known moderate to severe renal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Shalansky-Goldberg, MD, Principal Investigator — University of Pennsylvania; Pamela Grady, Ph.D, Study Director — Boston Scientific Corporation
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Shlansky-Goldberg RD, Rosen MA, Mondschein JI, Stavropoulos SW, Trerotola SO, Diaz-Cartelle J. Comparison of polyvinyl alcohol microspheres and tris-acryl gelatin microspheres for uterine fibroid embolization: results of a single-center randomized study. J Vasc Interv Radiol. 2014 Jun;25(6):823-32. doi: 10.1016/j.jvir.2014.03.009. Epub 2014 Apr 29. PMID 24788209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants undergoing Uterine Fibroid Embolization for symptomatic uterine fibroids at the participating site, that met the study inclusion criteria, were approached for consent for inclusion into the study. Enrollment occurred from February 2006 to December 2009.
Groups:
- Contour SE Microspheres: Polyvinyl alcohol Microsphere embolization devices intended to provide targeted vascular occlusion or reduction of blood flow upon selective placement and are currently marketed for use in hypervascular tumors, including leiomyoma uteri and arteriovenous malformations
- Embosphere Microspheres: Biocompatible, hydrophilic, nonresorbable, microspheres used in the embolization of arteriovenous malformations, hypervascular tumors, and symptomatic uterine fibroids.
Period: Overall Study
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Started | 30 | 30
Completed | 27 | 29
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contour SE Microspheres | Embosphere Microspheres | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.9 (5) | 41.7 (5.4) | 42.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 18 | 39
  Unknown or Not Reported | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Two participants in the Embosphere group had missing values for Race.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 21 | 20 | 41
    White | 7 | 6 | 13
    More than one race | 0 | 2 | 2
    Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Previous or concurrent gynecological disease(s) [Number; unit: partcipants]
  # of participants with concurrent gyneco disease | 5 | 7 | 12
  # of participants without concurrent gyneco diseas | 25 | 23 | 48
Fibroid Related Symptoms [Number; unit: particpants] — Fibroid related symptoms is collected on the baseline CRF. A participant may have multiple symptoms present, thus the number may not add up to 30 per group or 60 total. The analysis indicates the number of participants with each symptom, thus the sum for all categories in the arm/group does not equal the overall number of participants in the group.
  particpants
    Abnormal Bleeding | 28 | 27 | 55
    Bulk/pressure | 20 | 25 | 45
    Pelvic Pain | 22 | 23 | 45
    Other | 8 | 10 | 18
Number of fibroids present greater than 2cm [Number; unit: particpants]
  0 fibroids | 1 | 0 | 1
  1 fibroid | 1 | 3 | 4
  2 fibroids | 2 | 5 | 7
  3 fibroids | 10 | 4 | 14
  4 fibroids | 2 | 2 | 4
  5 fibroids | 2 | 2 | 4
  6 fibroids | 3 | 2 | 5
  7-10 fibroids | 6 | 5 | 11
  >10 fibroids | 3 | 7 | 10
Number of fibroids present less than 2 cm [Number; unit: participants]
  0 fibroids | 3 | 3 | 6
  1 fibroid | 2 | 3 | 5
  2 fibroids | 2 | 1 | 3
  3 fibroids | 3 | 1 | 4
  4 fibroids | 4 | 2 | 6
  5 fibroids | 2 | 4 | 6
  6 fibroids | 3 | 3 | 6
  7-10 fibroids | 4 | 4 | 8
  >10 fibroids | 7 | 9 | 16
Type of fibroid present [Number; unit: participants] — The type of fibroid present is determined from the baseline MRI. A participant may have more than one type of fibroid present, thus the number may not add up to 30 per group or 60 total. The analysis indicates the number of participants with each type of fibroid, thus the sum for all categories in the arm/group does not equal the overall number of participants in the group.
  participants
    Submucosal | 16 | 20 | 36
    Subserosal | 26 | 24 | 50
    Intramural | 28 | 28 | 56
    Transmural | 14 | 17 | 31
    Other, specify | 0 | 0 | 0
    Cannot determine | 0 | 0 | 0
Dominant fibroid volume [Mean (Standard Deviation); unit: cm^3] | 203.3 (275.1) | 141.1 (179.6) | 172.2 (232.5)
Uterine Volume [Mean (Standard Deviation); unit: cm^3] | 1536.7 (937.3) | 1491.6 (1456.5) | 1514.2 (1214.5)
Maximal thickness of junctional zone [Mean (Standard Deviation); unit: mm] | 11.4 (6.6) | 10.9 (7.9) | 11.2 (7.2)
Maximal thickness of the endometrium [Mean (Standard Deviation); unit: mm] | 7.3 (2.8) | 8.9 (3.3) | 8.1 (3.2)
Minimal thickness of the myometrium [Mean (Standard Deviation); unit: mm] | 11.2 (5.1) | 9.5 (4.2) | 10.3 (4.7)
Concomitant adenomyosis [Number; unit: participants] — This measure contains the number of subjects with concomitant adenomyosis. If concomitant adenomyosis was noted, it was further classified as focal or diffuse.
  Not all subjects had concomitant adenomyosis noted. The sum for all categories in the arm/group does not equal the overall number of participants in the group, because the value only indicates if the measure was present.
  participants
    Focal | 7 | 5 | 12
    Diffuse | 2 | 2 | 4
    Cannot Determine | 0 | 0 | 0
Presence of endometrial scar [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 30 | 30 | 60
Presence of myometrial scar [Number; unit: participants]
  Yes | 7 | 7 | 14
  No | 23 | 23 | 46
Assessment of myometrial perfusion [Number; unit: participants]
  Normal | 30 | 28 | 58
  Mildly Decreased | 0 | 1 | 1
  Moderately Decreased | 0 | 0 | 0
  Severly Decreased/Infarcted | 0 | 0 | 0
Ovaries seen [Number; unit: participants]
  Yes | 29 | 29 | 58
  No | 1 | 1 | 2
Adnexal Pathology [Number; unit: participants] — This measure contains the number of subjects with adnexal pathology noted. If adnexal pathology was noted, it was further classified to be endometrioma/endometriosis, cyst, or other.
  Not all subjects had adnexal pathology noted. The sum for all categories in the arm/group does not equal the overall number of participants in the group.
  participants
    Endometrioma/Endometriosis | 0 | 1 | 1
    Cyst | 3 | 2 | 5
    Other | 2 | 0 | 2
Obvious contribution to the uterine blood supply from the ovarian artery [Number; unit: participants]
  Yes | 0 | 1 | 1
  No | 30 | 29 | 59
Maximal Thickness of the myometrium [Mean (Standard Deviation); unit: mm] | 26.8 (8.1) | 25.0 (7.4) | 25.9 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fibroid Devascularization Measured by Contrast Enhanced Magnetic Resonance Imaging (MRI)
Description: MRI uses a large circular magnet and radio waves to generate signals from atoms in the body. These signals are used to construct images of internal structures. Injection of contrast through an IV is done during the test to enhance the view of the uterus. Contrast enhanced MRI was used as a test in this study to verify if blood supply to the fibroids was blocked or interrupted (devascularization).
Time Frame: 24-hours post study procedure
Measure: Number; unit: participants
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 29 | 30
participants | 29 | 29

2. Secondary Outcome: Visual Analog Scale (VAS) Maximum Level of Nausea
Description: Maximum level of nausea was measured using the Visual Analog Scale(VAS). The patient is presented with a picture of a straight line that is 0-10 cm long. The left side of the line (0 cm) represents 'no nausea' and the right side (10cm) of the line represents 'worst nausea imaginable'. The patient is asked to place a mark on the line that represents their level of nausea. For example, a reading of 10cm = worst nausea imaginable.
Time Frame: 24 hours after study procedure
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 30 | 30
cm | 5.5 (3) | 4.8 (3.2)

3. Secondary Outcome: Visual Analog Scale (VAS) Maximum Level of Pain
Description: Maximum level of pain was measured using the Visual Analog Scale(VAS). The patient is presented with a picture of a straight line that is 0-10 cm long. The left side of the line (0 cm) represents 'no pain' and the right side (10cm) of the line represents 'worst imaginable'. The patient is asked to place a mark on the line that represents their level of pain. For example, a reading of 10cm = worst imaginable pain.
Time Frame: 24 hours after study procedure
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 30 | 30
cm | 6.0 (2.9) | 5.6 (2.8)

4. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy is the method that provides real-time X ray imaging used for guiding a variety of diagnostic and interventional procedures. Fluoroscopy time is described as the amount of time the patient underwent fluoroscopy.
Time Frame: During the study procedure (measured in minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 30 | 30
minutes | 31.1 (19.4) | 24.9 (8.7)

5. Secondary Outcome: Procedure Time
Description: Procedure time is the time in minutes of the first arterial puncture to time of hemostasis (stopping bleeding)
Time Frame: During the study procedure (measured in minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 30 | 30
minutes | 102 (49.9) | 95.6 (39.6)

6. Secondary Outcome: Any Adverse Events That the Participant Experienced
Description: Summary of investigator reported adverse events and adverse device effects, including all serious adverse events and unanticipated adverse device effects. Adverse events were collected systematically, meaning they were collected during the participant's follow-up visit, during telephone contacts, or during medical record review.
Time Frame: During the hospitalization stay post UFE
Measure: Number; unit: events
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 30 | 30
events | 68 | 58

7. Secondary Outcome: Uterine Fibroid Symptom Quality of Life Questionaire (UFS-QOL) Score
Description: The UFS-QoL asks the subjects feelings and experiences regarding the impact of uterine fibroid symptoms and experiences during the previous 3 months.
  The scores are added and the final total scores range from 0-100. The lowest actual raw score=8, the highest raw score=40, the possible raw score range=32. A formula is then used to transform the value(actual raw score-lowest possible raw score divided by possible raw score range x100). Higher symptom score values are indicative of greater symptom severity or bother and lower scores indicate minimal symptom severity (high scores = bad)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 30 | 30
Scores on a scale | 64.2 (20.6) | 65.1 (20.3)

8. Secondary Outcome: Uterine Fibroid Symptom Quality of Life Questionaire (UFS-QOL) Score
Description: as for outcome 7
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 28 | 28
Scores on a scale | 16.3 (12.1) | 22.7 (20.5)

9. Secondary Outcome: Uterine Fibroid Symptom Quality of Life Questionaire (UFS-QOL) Score
Description: The UFS-QoL asks the subjects feelings and experiences regarding the impact of uterine fibroid symptoms and experiences during the previous 3 months.
  The scores are added and the final total scores range from 0-100.The lowest actual raw score=8, the highest raw score=40, the possible raw score range=32. A formula is then used to transform the value(actual raw score-lowest possible raw score divided by possible raw score range x100). Higher symptom score values are indicative of greater symptom severity or bother and lower scores indicate minimal symptom severity (high scores = bad).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 26 | 28
Scores on a scale | 18.0 (15.5) | 22.9 (17.8)

10. Secondary Outcome: Health Related Quality of Life (HRQL)Subscores
Description: The HRQL subscales (concern, activities, energy/mood, control, self-conscious, and sexual function were collected from the UFS-QoL.
  Each individual subscale is added. HRQL Total (sum of 6 subscales); lowest possible raw score = 29, highest possible raw score=145. A formula is used to transform the HRQL raw scores (Highest possible score-actual raw score divided by possible raw score range x 100). Higher scores are indicative of a better HRQL and lower scores indicate a worse HRQL (High=good). The value reported for this measure is the average of all participants scores.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 29 | 29
Scores on a scale | 42.1 (20.2) | 42.0 (23.7)

11. Secondary Outcome: Health Related Quality of Life Subscores
Description: as for outcome 10
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 28 | 28
Scores | 90.0 (13.1) | 90.0 (11.7)

12. Secondary Outcome: Health Related Quality of Life Subscores
Description: as for outcome 10
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Number analyzed (Participants) | 25 | 28
Scores on a scale | 89.8 (14.5) | 89.9 (11.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline, 24 hours post-procedure, 3 month follow-up, and 12 month follow-up.
Arm/Group | Contour SE Microspheres | Embosphere Microspheres
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/30
Other Adverse Events (participants affected / at risk) | 25/30 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contour SE Microspheres (N=30) | Embosphere Microspheres (N=30)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contour SE Microspheres (N=30) | Embosphere Microspheres (N=30)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (5)
Fatigue (General disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 3 (3) | 4 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 5 (5) | 6 (7)
Incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Vaginal Exfoliation (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vascular Injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Vasospasm (Vascular disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (14) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication to remove any confidential information or other proprietary information of Sponsor.